CLINICAL TRIAL: NCT01082003
Title: A Single Center, Prospective Treatment Trial to Assess Prophylactic Use of Trental (Pentoxifylline) and Vitamin E to Prevent Capsular Contracture After Implant Reconstruction in Patients Requiring Adjuvant Radiation Therapy
Brief Title: Prevention of Capsular Contracture Using Trental and Vitamin E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Legacy Health System (Other)
Responsible Party: Principal Investigator, Nathalie Johnson, Principal Investigator, Legacy Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LHS T-E01
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Capsular Contractures
Keywords: Capsular contractures in breast cancer patients
MeSH Terms: interventions — Pentoxifylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Permanent Implant (Other): Trental and Vitamin E for 6 months
  Interventions: Drug: Trental
- Tissue Expander (Other): Trental and Vitamin E for 6 months
  Interventions: Drug: Trental

INTERVENTIONS:
Drug: Trental — Trental (pentoxifylline) 400 milligrams three times a day in combination with vitamin E, 400 international units orally twice daily for six months.

SUMMARY:
The main purpose of this research study is to determine if the use of Trental and Vitamin E will decrease the incidence and severity of contractures (shrinking and or hardening of tissue surrounding the implant) associated with breast implant reconstruction following radiation treatment. Another goal is to find out the impact that Trental and Vitamin E have on implant loss or need for surgical intervention in the setting of chest wall radiation after reconstruction. In addition, the investigators want to evaluate the patient's sense of well being and quality of life.

DETAILED DESCRIPTION:
This is a single center, 18-month study in which 30 women will receive Trental (pentoxifylline) 400 milligrams three times a day in combination with vitamin E, 400 international units orally twice daily for six months. Subjects will begin the treatment regimen within four weeks after completion of radiation treatment and will remain on the study drugs for six months. Following completion of active treatment, all subjects will enter the twelve-month observational phase of the trial in which they will be evaluated for changes in breast tissue using the following objective tools: Bakers Grade Assessment, Visual Analog Scale (VAS), implant revision or loss, breast photographs, adverse event assessment and the Quality of Life tool (SF-12).

ELIGIBILITY:
Inclusion Criteria:

* Female subjects
* > 18 years of age
* Expected survival at least > 6 months
* Undergone mastectomy with expander or implant reconstruction > 3 weeks before radiation therapy
* Completed chest wall irradiation in the past two weeks
* Willing to stop herbal medications as directed by physician
* Willing to stop daily use of supplemental vitamin E (Multivitamin with vitamin E component is acceptable)
* Willing to travel to a Legacy Health System facility
* Agree to attend study visits outside of standard of care visits
* Normal PT-INR for subjects taking Coumadin

Exclusion Criteria:

* < 18 years of age
* Pregnant or lactating
* Have final implant placed < 3 weeks before start of radiation therapy
* Have evidence of ongoing infection or implant exposure before start of radiation therapy
* Radiation completed more than 16 days prior to study start
* Retinitis Pigmentosa
* Unable to comply with protocol
* Unable to provide written informed consent
* Unwilling or unable to stop supplemental vitamin E
* PT-INR outside of acceptable range for subjects taking Coumadin
* Investigator does not believe study participation, for any reason is in the best interest of the patient

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-10; Primary Completion 2013-08 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Measure number and grade of contractures occurring after implant reconstruction and radiation treatment in subjects receiving Trental and vitamin E combination compared to placebo using the Bakers grade assessment | 6 months

SECONDARY OUTCOMES:
Number of implant revisions or loss of implants due to post radiation changes in subject receiving Trental and vitamin E compared to placebo through patient interview with research staff | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Johnson, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Good Samaritan Medical Center, Portland, Oregon, United States